CLINICAL TRIAL: NCT03973580
Title: Altering High-risk Trajectories in Adolescent Anxiety Via Attention Bias Modification Training: Neural Predictors and Mechanisms (ABM Study)
Brief Title: Using Attention Training to Reduce Adolescents' Anxious Symptoms
Acronym: ABM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of the COVID-19 pandemic (Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention).
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Elizabeth Hayden, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Western HSREB #113928
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Attentional Bias; Anxiety
Keywords: Attentional Bias; Anxiety risk; Adolescence; Eye-tracking; Resting-state functional magnetic resonance imaging
MeSH Terms: conditions — Anxiety Disorders | interventions — potassium channel subfamily K member 3

STUDY DESIGN:
Intervention Model Description: Sixty adolescents will be randomly assigned to an active ABM task (n=30) or a control task (n=30) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomized assignment procedure will be conducted solely by the PI. All other research staff and participants will be blind to the assigned condition throughout the course of the study. The PI will use a random number generator in Excel to assign a number 1-10 for each participant. The number will be given to the study coordinator, who notes the number in the participant's file. Participants will be assessed by the coordinator or other research staff. The research staff goes to each participant's home to conduct the ABM training protocol, where the number noted in this participant's file will be entered at the start of the training task to assign the participant to either the ABM task or the control task. The PI will not run the tasks. In communicating with participants, the terms baseline, outcome, and training will not be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attentional Bias Modification (ABM) group (Active Comparator): Participants in this arm will participate in a six-session ABM task, one session per week.
  Interventions: Behavioral: Attentional Bias Modification (ABM) task
- Control group (Placebo Comparator): Participants in this arm will participate in a six-session control task, one session per week.
  Interventions: Behavioral: Control task

INTERVENTIONS:
Behavioral: Attentional Bias Modification (ABM) task — Participants will be presented with a fixation cross (500ms) followed by a pair of identity-matched, angry-neutral faces (1000ms). The pair presentation is replaced by a single arrow-probe (1000ms) in the position of the neural face. Inter-trial intervals (ITI) are 500ms. Participants indicate arrow direction (left or right) by pressing one of two buttons as quickly as possible. By responding to the probe that always replaces the neutral face, participants learn to attend to the non-threat cues and away from threat cues. There are 120 trials of angry-neutral faces in total, and 40 other catch trials with neutral-neutral faces.
  Arms: Attentional Bias Modification (ABM) group
Behavioral: Control task — The control task is identical with the ABM task, except that in the 120 angry-neutral trials, the arrow-probe replaces the angry face and the neutral face with equal probabilities (60 trials each).
  Arms: Control group

SUMMARY:
During adolescence, youth undergo rapid developmental change and in some cases experience increases in worries and fearfulness, although the mechanisms that underlie this change are unclear. Previous studies indicate that heightened Attentional Bias (AB) toward threat-related cues may increase fearfulness, and it may be possible to change AB using a computerized, Attention Bias Modification task (ABM). This study will recruit healthy youth with elevated anxious symptoms to index attentional tendencies toward threat-related stimuli using cutting-edge techniques, and to test the effect of a computerized attention training task in altering attention to threatening cues. The investigators will also examine the role of ABM in changing youth's attention-related resting-state functional connectivity (rsFC), a neural marker of at-rest cognition.

DETAILED DESCRIPTION:
Adolescence is a critical period for increases in anxious symptoms, potentially due to etiologically significant Attention Biases (AB) favoring threatening cues. However, the specific facets of AB that drive this vulnerability as well as their neurocognitive correlates are unclear, due in large part to the poor psychometric properties of the traditional assessment of AB in this field. By using both a standard behavioral task and a novel eye-tracking task, this study aims to unpack the nuanced facets of AB related to anxiety risks. Additionally, well-controlled Attentional Bias Modification (ABM) tasks designed to train attention away from threatening cues can be used to experimentally manipulate the causal mechanisms of interest, and to test whether ABM reduces symptoms and alters patterns of resting-state functional connectivity (rsFC, the intrinsic brain activity that occurs outside specific tasks) that characterize anxiety risks.

This study will recruit 60 11-13-year-old healthy adolescents with heightened anxious symptoms but without clinically significant anxiety disorders. They will be randomized to a six-session ABM training or a placebo task. Both before and after the training, the investigators will assess their anxious symptoms, AB, and rsFC. By examining the risk processes prior to the onset of clinically significant anxiety disorders, our work will make important new contributions to our understanding of how AB eventuates in anxiety and will have direct implications for early identification of youth at highest risk for anxiety disorders, and the targets that should be focused on in preventative efforts.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking 11-13-year-old youth without significant medical, psychological, cognitive, or language impairments.

Exclusion Criteria:

* Adolescents with clinically significant anxiety disorders or conditions in conflict with MRI scanning (e.g., orthodontics) will be excluded.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent-reported anxious symptoms at 3 weeks follow-up | 3 weeks from baseline (after completing the 3rd weekly training session)
  Parent-reported anxious symptoms will be assessed by the Child Behavior Checklist questionnaire. The anxious syndrome subscale will be used with a score summed across the 12 items of this subscale. Scores for each item range from 0 to 2, and scores for the subscale range from 0 to 24. Higher scores indicate greater anxious symptoms.
Change from baseline in parent-reported anxious symptoms at 6 weeks follow-up | 6 weeks from baseline (after completing the 6th weekly training session)
  Parent-reported anxious symptoms will be assessed by the Child Behavior Checklist questionnaire. The anxious syndrome subscale will be used with a score summed across the 12 items of this subscale. Scores for each item range from 0 to 2, and scores for the subscale range from 0 to 24. Higher scores indicate greater anxious symptoms.
Change from baseline in youth self-reported anxious symptoms at 3 weeks follow-up | 3 weeks from baseline (after completing the 3rd weekly training session)
  Youth self-reported anxious symptoms will be assessed by the Youth Self Report questionnaire. The anxious syndrome subscale will be used with a score summed across the 12 items of this subscale. Scores for each item range from 0 to 2, and scores for the subscale range from 0 to 24. Higher scores indicate greater anxious symptoms.
Change from baseline in youth self-reported anxious symptoms at 6 weeks follow-up | 6 weeks from baseline (after completing the 6th weekly training session)
  Youth self-reported anxious symptoms will be assessed by the Youth Self Report questionnaire. The anxious syndrome subscale will be used with a score summed across the 12 items of this subscale. Scores for each item range from 0 to 2, and scores for the subscale range from 0 to 24. Higher scores indicate greater anxious symptoms.

SECONDARY OUTCOMES:
Change from baseline in response-time-indexed Attentional Bias (AB) at 6 weeks follow-up | 6 weeks from baseline (after completing the 6th weekly training session)
  This outcome will be assessed by a behavioral dot-probe task.
Change from baseline in eye-movement-indexed Attentional Bias (AB) at 6 weeks follow-up | 6 weeks from baseline (after completing the 6th weekly training session)
  This outcome will be assessed by an eye-tracking task.
Change from baseline in resting-state functional connectivity (rsFC) | 6 weeks from baseline (after completing the 6th weekly training session)
  rsFC will be assessed by resting-state functional magnetic resonance imaging (fMRI).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Hayden, Ph.D, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the PI. Requests with the sole purpose of research will be approved. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Sanchez A, Romero N, De Raedt R. Depression-related difficulties disengaging from negative faces are associated with sustained attention to negative feedback during social evaluation and predict stress recovery. PLoS One. 2017 Mar 31;12(3):e0175040. doi: 10.1371/journal.pone.0175040. eCollection 2017. PMID 28362826
- [Result] Beard C, Sawyer AT, Hofmann SG. Efficacy of attention bias modification using threat and appetitive stimuli: a meta-analytic review. Behav Ther. 2012 Dec;43(4):724-40. doi: 10.1016/j.beth.2012.01.002. Epub 2012 Jan 18. PMID 23046776
- [Result] Bar-Haim Y, Lamy D, Pergamin L, Bakermans-Kranenburg MJ, van IJzendoorn MH. Threat-related attentional bias in anxious and nonanxious individuals: a meta-analytic study. Psychol Bull. 2007 Jan;133(1):1-24. doi: 10.1037/0033-2909.133.1.1. PMID 17201568
- [Result] Liu P, Taber-Thomas BC, Fu X, Perez-Edgar KE. Biobehavioral Markers of Attention Bias Modification in Temperamental Risk for Anxiety: A Randomized Control Trial. J Am Acad Child Adolesc Psychiatry. 2018 Feb;57(2):103-110. doi: 10.1016/j.jaac.2017.11.016. Epub 2017 Nov 28. PMID 29413142